CLINICAL TRIAL: NCT01450488
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Activity of Oral AB1010 Administered at 2 Dose Levels to Patients With Primary Progressive or Relapse-free Secondary Progressive Multiple Sclerosis
Brief Title: Masitinib in Primary Progressive Multiple Sclerosis or Relapse-free Secondary Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB04011
Record Dates: First submitted 2011-10-06; First posted 2011-10-12 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Multiple Sclerosis
Keywords: primary progressive multiple sclerosis; relapse-free secondary progressive multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — masitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- masitinib 3 mg/kg/day (Experimental)
  Interventions: Drug: masitinib
- masitinib 6 mg/kg/day (Experimental)
  Interventions: Drug: masitinib

INTERVENTIONS:
Drug: masitinib — masitinib 3 mg/kg/day
  Arms: masitinib 3 mg/kg/day
Drug: masitinib — masitinib 6 mg/kg/day
  Arms: masitinib 6 mg/kg/day

SUMMARY:
The purpose of this study is to evaluate the activity of oral AB1010, administered at two dose levels during 3 years to patients with primary or secondary progressive multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 60 years, from both sex, and suffering from multiple sclerosis either primary progressive or secondary progressive without relapse within 2 years before inclusion.
2. Patients with EDSS score in the range of 2 to 6.5, inclusive
3. EDSS progression ≥ 1 point within 2 years before inclusion

Exclusion Criteria:

1. Disease other than MS responsible for clinical signs and/or MRI lesions
2. Secondary progressive MS with relapse in the 2 years before inclusion
3. Treatment with interferon or glatiramer acetate within four weeks prior to treatment allocation
4. Treatment with oral or systemic corticosteroids or ACTH within four weeks prior to treatment allocation.
5. Active current bacterial, viral (including hepatitis B and C, HIV, EBV, CMV, herpes zoster, herpes simplex), fungal, mycobacterium, protozoan, or other infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2005-06; Primary Completion 2007-07 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
change in MSFC | 12 months
  average change in multiple sclerosis functional composite (MSFC) score relative to baseline, with clinical response defined as a > 100% improvement (increase) from baseline

SECONDARY OUTCOMES:
MSFC subcategories | 12 months
  timed 25-foot walk (T25FW)
Expanded Disability Status Scale (EDSS) | 12 months
MFSC subcategories | 12 months
  9-Hole Peg Test (9-HPT)
MFSC subcategories | 12 months
  Paced Auditory Addition Test (PASAT-3'')

REFERENCES:
- [Result] Vermersch P, Benrabah R, Schmidt N, Zephir H, Clavelou P, Vongsouthi C, Dubreuil P, Moussy A, Hermine O. Masitinib treatment in patients with progressive multiple sclerosis: a randomized pilot study. BMC Neurol. 2012 Jun 12;12:36. doi: 10.1186/1471-2377-12-36. PMID 22691628
- See also: Link to article — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3467179/